CLINICAL TRIAL: NCT04047550
Title: Respiratory Control and Prevention of Opioid-Induced Respiratory Depression After Surgery
Brief Title: Respiratory Control and Narcotic Effects
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00046973
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Ventilatory Depression; Opioid Intoxication; Opioid Toxicity
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Ventilatory chemosensitivity — Using this technique, the patient first voluntarily hyperventilates to a PETCO2 value of 20-25 mmHg, then undergoes a rebreathing test allowing the PCO2 to rise to 55-60 mmHg while PETO2 is maintained at 150 mmHg. The procedure is then repeated with PETO2 clamped at 50 mmHg. Parameters derived from this method include slopes of the ventilatory response during hyperoxia and hypoxia.

SUMMARY:
The aim of this study is to provide data that will assess the role of ventilatory chemosensitivity (respiratory drive) in determining postoperative respiratory depression due to opioids. In a group of patients requiring surgery and admission to hospital, before surgery, ventilatory chemosensitivity will be assessed in the presence or absence of an infusion of remifentanil. Parameters will be correlated with ventilatory depression events after surgery. A secondary aim is to determine whether respiratory depression is more likely during specific phases of sleep.

DETAILED DESCRIPTION:
The study aims to test the following hypotheses:

Low respiratory drive is predictive of opioid-induced respiratory depression as defined by end-tidal PCO2 (PETCO2) >50 mmHg, ventilation <20% below baseline or pulse oximeter reading (SpO2) <90%.

Respiratory depression is more likely during certain sleep stages, specifically slow wave sleep.

Respiratory Drive. Before surgery each patient's hypercapnic ventilatory response under conditions of mild hypoxia and mild hyperoxia. Using this technique, the patient first voluntarily hyperventilates to a PETCO2 value of 20-25 mmHg, then undergoes a rebreathing test allowing the PCO2 to rise to 55-60 mmHg while end-tidal PO2 (PETO2) is maintained at 150 mmHg. The procedure is then repeated with PETO2 clamped at 50 mmHg. Parameters derived from this method include slopes of the ventilatory response during hyperoxia and hypoxia. The slope during mild hypoxia is felt to be an index of peripheral chemoreceptor function, while the hyperoxic slope is more indicative of central respiratory drive.

These two maneuvers will then be repeated during an infusion of the ultra-short acting opioid, remifentanil. Remifentanil will be administered to achieve a specified effect site concentration selected to produce a 30% decrease in ventilation using a standard pharmacokinetic model implemented on a widely-used shareware program (TIVATrainer, www.eurosaver.eu). Recovery from ventilatory depression occurs within 10 minutes of discontinuation of the infusion.

Sleep Test. During a night before surgery a sleep test based on peripheral arterial tone will be performed at home (WatchPAT™, Itamar Medical, Franklin, MA) and will provide a formal measure of obstructive sleep apnea. This test requires only a device mounted on a finger that assesses SpO2 and peripheral tone, and an accelerometer on the chest to assess breathing movements. Respiratory indices calculated using this technology correlates with those calculated from standard polysomnography. The same testing will be used postoperatively from the time the patient enters the post anesthesia care unit (PACU) until the following morning. Recording of the same variables will then continue: inter-breath interval, respiratory minute volume (using an electrical impedance device: ExSpiron™, Respiratory Motion, Waltham, MA), abdominal strain gauge recording, transcutaneous PCO2 (SenTec, Fenton, MO), and sleep measures. The data stream will then be divided into 5 minute epochs. During each epoch the sleep state (awake, stages 1-4 slow wave sleep, rapid eye movement (REM) sleep), opioid consumption, respiratory variables and apnea/hypopnea index (AHI) will be assessed. Subjects will have the option to opt in or out of participation in the overnight sleep study.

Long-Term Pulse Oximetry. For the entire postoperative period until discharge we will record opioid consumption and SpO2/heart rate using a wrist oximeter (WristOx™, Nonin Medical, Plymouth, MN).

Postoperative parameters of respiratory depression include hypercapnia (transcutaneous PCO2), hypoxemia, apneas, low respiratory minute volume and sleep state.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older, undergoing major abdominal or urological surgery requiring at least one overnight hospital stay

Exclusion Criteria:

Pregnancy Adverse reaction to remifentanil Opioid-use within the past month Dependency on supplemental oxygen Brain injury in the past year Coronary artery disease Sickle cell disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery requiring opioids for postoperative analgesia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Opioid related respiratory depression (OIRD) frequency | From the arrival of the patient in the post anesthesia care unit until the first postoperative morning
  A respiratory event is defined as one or more of the following:
  1. Respiratory rate <60% of baseline
  2. Minute ventilation (MV) <60% of predicted value based on body surface area (BSA). Predicted MV for men=4 x BSA, for women=3.5 x BSA
  3. Pulse oximeter reading (SpO2) <90% (breathing room air) or <92% (breathing supplemental O2)
  4. Transcutaneous PCO2 >50 mmHg
  5. Central or obstructive apnea/hypopnea detected by WatchPAT (Itamar Medical, Atlanta, GA) based on decrease in peripheral arterial tone amplitude, increase in heart rate and decrease in SpO2 ≥3% or snoring in the absence of body movement.
  Events must last 1 minute or more to be counted. Events occurring within one minute of each are combined as a single event.

SECONDARY OUTCOMES:
Frequency of OIRD during specific sleep stages | From the arrival of the patient in the post anesthesia care unit until the first postoperative morning
  OIRD as defined in the primary outcome, as a function of sleep stage postoperatively, as measured using the WatchPAT™ (Itamar Medical, Franklin, MA)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Moon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No